CLINICAL TRIAL: NCT07327073
Title: The Effect of High-intensity Intermittent Exercise and Moderate-intensity Continuous Exercise on Serum Irisin Levels, Disease Activity, Functional Status, and Quality of Life in Patients With Axial Spondyloarthritis: a Prospective, Randomized Study
Brief Title: The Effect of Exercise on Serum Irisin Levels and Clinical Parameters in Patients With Axial Spondyloarthritis.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Collaborators: Scientific Research Projects (Unknown)
Responsible Party: Principal Investigator, Nazife Kapan, Asst. Prof., Kirsehir Ahi Evran Universitesi
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AhiEvranU-FTR-NK-AS
Record Dates: First submitted 2025-12-25; First posted 2026-01-08 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Ankylosing Spondylitis (AS); Irisin
Keywords: ankylosing spondylitis; exercise; irisin
MeSH Terms: conditions — Spondylitis, Ankylosing; Motor Activity | interventions — High-Intensity Interval Training; Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- high-intensity exercise (Experimental): Patients in this group will receive information and education about their condition and will be instructed to continue their current medical treatment and attend follow-up appointments regularly. Additionally, this group will undergo a high-intensity interval training (HIIT) program with a physiotherapist for 40 sessions in total, 5 sessions per week for 8 weeks, each lasting 35 minutes. Patients will work at 80% to 100% of their maximum heart rate. The first 4 weeks will be at 80% of maximum heart rate, followed by 85%, 90%, 95%, and finally 100%. This protocol will consist of 4 active periods of 4 minutes each at 80% to 100% of maximum heart rate (percentage to be determined weekly) and 3 rest periods of 3 minutes each at 60-70% of maximum heart rate (4x4 minutes). Each session will include a 5-minute warm-up before HIIT and a 5-minute cool-down after HIIT, for a total exercise time of 35 minutes.
  Interventions: Other: High-Intensity Interval Training
- moderate intensity exercise (Experimental): Patients in this group will receive information and education about their condition and will be instructed to continue their current medical treatment and attend regular follow-up appointments. Additionally, these patients will undergo a 40-minute, 5-session, 40-minute moderate-intensity continuous exercise (MCIT) program with a physiotherapist over 8 weeks. Patients will exercise at 50-70% of their maximum heart rate and with an RPE of 11-13 for 30 minutes. Each session will include a 5-minute warm-up before MCIT and a 5-minute cool-down after MCIT, for a total exercise duration of 40 minutes.
  Interventions: Other: Moderate-Intensity Continuous Exercise
- control (Active Comparator): Patients in this group will receive information and education about their illness and will be advised to continue their current medical treatment and attend their follow-up appointments regularly.
  Interventions: Other: control group

INTERVENTIONS:
Other: High-Intensity Interval Training — Patients will be trained at 80% to 100% of their maximum heart rate. For the first 4 weeks, they will train at 80% of their maximum heart rate, then at 85%, 90%, 95%, and finally 100%. This protocol will consist of 4 active periods of 4 minutes each at 80% to 100% of maximum heart rate (percentage to be determined weekly) and 3 rest periods of 3 minutes each at 60-70% of maximum heart rate (4x4 minutes). Each session will include a 5-minute warm-up before HIIT and a 5-minute cool-down after HIIT, for a total exercise time of 35 minutes.
  Arms: high-intensity exercise
Other: Moderate-Intensity Continuous Exercise — Patients will be trained for 30 minutes at 50% to 70% of their maximum heart rate and with an RPE of 11-13. Each session will include a 5-minute warm-up before MCIT and a 5-minute cool-down after MCIT, for a total exercise time of 40 minutes.
  Arms: moderate intensity exercise
Other: control group — They will be given information and education about their illnesses and will be advised to continue their current medical treatment and attend their follow-up appointments regularly.
  Arms: control

SUMMARY:
This study aimed to investigate the effects of high-intensity intermittent exercise and moderate-intensity continuous exercise on serum irisin levels, disease activity, functional status, and quality of life in patients with axial spondyloarthritis.

DETAILED DESCRIPTION:
Axial spondyloarthritis (axSpA) is a chronic inflammatory rheumatic disease affecting young individuals, with a prevalence of 0.3-1.4%. The main features of the disease include inflammatory back pain, reduced joint mobility, and functional disability. In addition, accumulating evidence over recent years has demonstrated that inflammatory rheumatic diseases are associated with an increased risk of cardiovascular disease. Exercise constitutes an important component of the management of inflammatory rheumatic diseases and is widely used to reduce pain and improve joint mobility.

Irisin is a myokine secreted by skeletal muscle through the cleavage of the membrane protein fibronectin type III domain-containing protein 5 (FNDC-5). Irisin is considered a mediator of exercise-induced metabolic benefits and has been shown to exert protective effects in several non-metabolic diseases. At the molecular level, irisin contributes to increased energy expenditure and metabolic regulation by promoting the browning of white adipose tissue. Previous studies have demonstrated that serum irisin levels increase following exercise.

Studies evaluating the role of irisin in ankylosing spondylitis have reported lower serum irisin levels in patients with more severe disease manifestations. However, no studies investigating the effects of exercise therapy on serum irisin levels in patients with axial spondyloarthritis have been identified in the literature. Previous research has focused on the relationship between disease severity and serum irisin levels, as well as the association between serum irisin levels and cardiovascular disease in patients with ankylosing spondylitis. Overall, low serum irisin levels are thought to be indicative of subclinical atherosclerosis, increased cardiovascular risk, and more severe disease. Evaluating the relationship between serum irisin levels and exercise in patients with axial spondyloarthritis may provide important contributions to disease management and follow-up. Therefore, the present study aimed to investigate the effects of high-intensity intermittent exercise and moderate-intensity continuous exercise on serum irisin levels, disease activity, functional status, and quality of life in patients with axial spondyloarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with axillary spondyloarthropathy according to ASAS diagnostic criteria,
* Having a high disease severity (ASDAS-CRP above 2.1),
* Being sedentary (not engaging in physical activity at least 3 days a week in the last 3 months),
* Having no change in ankylosing spondylitis medical treatment in the last 3 months,
* Not having any orthopedic, neurological, cardiovascular, or mental disease that would affect exercise,
* Not using any assistive devices for ambulation,
* Having a BMI of 25 kg/m2 or less,
* Male and female patients aged 18-50 years.

Exclusion Criteria:

* Those with uncontrolled cardiopulmonary disease (such as hypertension, chronic obstructive pulmonary disease, heart failure),
* Having comorbidities that reduce exercise capacity,
* Pregnancy,
* Malignancy,
* Those with a recent history of surgery,
* Those who have engaged in regular exercise (aquatic exercise, land exercise, etc.) in the previous 3 months

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
serum irisin level | Before treatment and after treatment (week 8)
  Blood samples will be taken from patients one day before the start of treatment, after a 12-hour fast, and again the morning after a 12-hour fast, immediately after the end of treatment. The collected blood samples will be centrifuged at 1500 g for 10 minutes to obtain serum. The obtained serum will be stored at -80°C until the day of the study. The aim of these serum samples is to determine the level of irisin.

SECONDARY OUTCOMES:
Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | Before treatment, after treatment (week 8)
  The BASDAI score consists of 6 questions. Patients are asked to rate each question on a scale of 0 to 10, based on their symptoms one week prior, with 'none' receiving 0 points and 'very severe' receiving 10 points. The scores from questions 5 and 6 are then added together, divided by 2, and added to the other scores. The total is then divided by 5 to obtain the BASDAI score. A BASDAI score of 4 or higher indicates that the disease is out of control and that the patient's treatment, particularly biological agents, should be reviewed. To assess treatment response, a 50% improvement in the BASDAI score or at least a 2-unit reduction on a 10-point scale is required.
Ankylosing Spondylitis Activity Scoring-CRP (ASDAS-CRP) | Before treatment, after treatment (week 8)
  The ASDAS score is a combined scoring system that measures disease activity. It is calculated by adding the CRP value to clinical findings. Based on the resulting score, disease activity is grouped as inactive, low, high, and very high. For evaluation to initiate biological therapy, the ASDAS score must be at least 2.1. A change of 1.1 or higher in the ASDAS score is considered a significant improvement, while changes of 2.0 or higher are considered major improvements. A change of 0.9 or higher in the ASDAS score is required for a disease activity flare-up.
Bath Ankylosing Spondylitis Functional Index (BASFI) | Before treatment, after treatment (week 8)
  Patients are asked a total of 10 questions, including functional questions, and are asked to rate each question between 0 and 10, with 0 points for 'easy' and 10 points for 'impossible'. The points given for each question are added together and divided by 10 to obtain the BASFI score.
Bath Ankylosing Spondylitis Metrology Index (BASMI) | Before treatment, after treatment (week 8)
  Metrological evaluations of patients are performed using this scoring system. The score is calculated by measuring lumbar lateral flexion, tragus wall distance, modified Schober test, cervical rotation, and intermalleolar distance. It is used as a follow-up parameter in spinal mobility measurements.
Ankylosing Spondylitis Quality of Life Scale (ASQoL) | Before treatment, after treatment (week 8)
  The system consists of 18 questions, where "yes" is worth 1 point and "no" is worth 0 points. Points are added up to calculate the score. A higher score indicates a poorer quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Kırşehir Ahi Evran Üniversitesi, Kırşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No